CLINICAL TRIAL: NCT03222765
Title: Early Prevention of Diabetes Complications in People With Hyperglycaemia in Europe: e-PREDICE Study
Brief Title: Prevention of Microvascular Complications in Prediabetes e-PREDICE Study
Acronym: ePREDICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Evidem Consultores SL (Industry)
Collaborators: European Commission (Other); Boehringer Ingelheim (Industry); Merck Serono International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EU-FP7 279074
Record Dates: First submitted 2017-06-20; First posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-06

CONDITIONS: PreDiabetes
Keywords: prediabetes lifestyle drugs microvascular complications
MeSH Terms: conditions — Prediabetic State | interventions — Metformin; Linagliptin

STUDY DESIGN:
Intervention Model Description: Randomized, parallel , single-blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Two groups (linagliptin vs placebo) double-blind Two groups (metformin & metformin+linagliptin) single-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): * Placebo
  * Lifestyle modification (diet and physical activity recommendations)
  Interventions: Drug: Placebo, metformin, linagliptin, linagliptin + metformin
- Metformin (Experimental): * Metformin
  * Lifestyle modification (diet and physical activity recommendations)
  Interventions: Drug: Placebo, metformin, linagliptin, linagliptin + metformin
- Linagliptin (Experimental): * Linagliptin
  * Lifestyle modification (diet and physical activity recommendations)
  Interventions: Drug: Placebo, metformin, linagliptin, linagliptin + metformin
- Linagliptin and Metformin (Experimental): * Fixed dose combination of Linagliptin and metformin
  * Lifestyle modification (diet and physical activity recommendations)
  Interventions: Drug: Placebo, metformin, linagliptin, linagliptin + metformin

INTERVENTIONS:
Drug: Placebo, metformin, linagliptin, linagliptin + metformin

SUMMARY:
Background: A significant proportion of pre-diabetics, show macro and micro vascular complications associated with hyperglycaemia. Although many trials have demonstrated the efficacy of lifestyle and pharmaceutical interventions in diabetes prevention, no trial has evaluated the extent to which mid- and long-term complications can be prevented by early interventions on hyperglycaemia.

Aims: To assess the long-term effects on multiple complications of hyperglycaemia of early intensive management of hyperglycaemia with linagliptin, metformin or their combination added to lifestyle intervention (LSI) (diet and physical activity), compared with LSI alone in adults with non-diabetic intermediate hyperglycaemia (IFG, IGT or both).

Study Design: Investigator initiated (non-commercial), long-term, multi-centre, randomised, partially double blinded, placebo controlled, phase-IIIb clinical trial with prospective blinded outcome evaluation. Participants will be randomised to four parallel arms: 1) LSI + 2 placebo tablets/day; 2) LSI + 2 Metformin tablets of 850 mg/day; 3) LSI + 1 Linagliptin tablets of 5 mg/day and 1 placebo; 4) LSI + 2 tablets of a fixed-dose combination of Linagliptin 2.5mg and Metformin 850 /day. Active intervention will last for at least 2 years.

Setting and population: Males and Females with pre-diabetes (IFG, IGT or both) aged 45 to 74 years selected from primary care screening programs in 14 clinical centres from 10 countries: Australia, Austria, Bulgaria, Greece, Italy, Kuwait, Poland, Serbia, Spain and Turkey and . (N=1000)

Main Outcomes: The primary endpoint is a combined continous variable: "the microvascular complication índex" (MCI) composed by a linear combination of the Early Treatment Diabetic Retinopathy Study Scale (ETDRS) score (based on retinograms), the level of urinary albumin to creatinine ratio, and a measure of distal small fibre neuropathy (sudomotor test by SUDOSCAN), measured during baseline visit and at 24th and 48th month visits after randomisation. In addition, serological biomarkers of inflammation, vascular damage, non-alcoholic fatty liver disease, insulin secretion, measures of quality of life, sleep quality, neuropsychological evaluation and endothelial function will be also evaluated in a subset of participants.

ELIGIBILITY:
Inclusion criteria

* Impaired Fasting Glucose (IFG): Fasting Plasma Glucose (FPG) 6.1 to 6.9mmol/l and 2-hour Plasma Glucose (2-h PG): <7.8mmol/L;
* Impaired Glucose Tolerance (IGT): FPG <7.0mmol/L and 2h PG >_7.8 and <11.1 mmol/L -Informed consent given

Exclusion Criteria:

* Type 1 diabetes (T1D)
* known or screen-detected Type 2 diabetes (T2D).
* Use of any anti-diabetic drug within the 3 months prior to inclusion.
* Previous cardiovascular event, stroke or revascularization procedure of any arterial territory
* Morbid obesity (BMI>45)
* Current renal replacement therapy.
* Renal function impairment: GFR <60 ml/min/1.73m2.
* Previous diagnosis of liver cirrhosis or chronic hepatitis
* Elevation of liver enzymes (AST/AST) >3 times of the upper normal ranges** (6m or BL).
* Previous diagnosis of acute or chronic pancreatitis
* Elevation of pancreatic enzymes (Amylase/Lipase) >3 times of the upper normal ranges (6m or BL).
* Previous diagnosis of Chronic Heart Failure (NYHA class III or higher).
* Organ transplant or waiting for organ transplant.
* Diagnosis of malignant neoplasm requiring chemotherapy, surgery, radiation or palliative therapy in the previous 5 years.
* End-stage or metastatic cancer.
* Known or suspected hypersensitivity to trial products or related products.
* Known use of non prescribed narcotics or illicit drugs.
* Simultaneous participation in any other clinical trial of an investigational agent.
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant.
* Cataract that impedes the retinal evaluation of both eyes.
* Ocular surgery planned in the next 6 months
* Concomitant intraocular treatment (retina or choroid).
* Tropicamide allergy
* Participants with screen retinogram not optimal for retinal assessment
* Complete amputation of one/ both hands or one/both feet.
* Dementia, mental disorder or evident cognitive impairment unable to give informed consent.
* Institutionalization (nursing/mental health home, hospital, prison, etc).
* Suspected renal artery stenosis Recent gastrointestinal bleeding (within the last year)
* Any circumstance where ongoing medication might lead to potential adverse drug effect.
* Any other acute condition or exacerbation of chronic condition that in the investigator's opinion would interfere with the trial initiation or visit schedules or procedures.

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2015-03-15 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Microvascular Complication Index "MIC" : | 2-year
  linear combination of three continous variables: ETRSD score, UACR and sudomotor index
Diabetic Retinopathy: Scale ETDRS | 2-year
  ETDRS Score
Urine albumin to creatinine ratio (UACR) | 2-year
  Ratio albumin to creatinine in mg/dl
Sudomotor Index | 2-year
  SUDOSCAN sweat function

SECONDARY OUTCOMES:
incidence of diabetes | 2-year
  new cases of Type 2 Diabetes
endothelial dysfunction | 2-year
  ENDOPATH measurement
Insulin sensitivity | 2-year
  Insulin secretion and beta-cell function
Inflammation biomarkers | 2-years
NAFLD biomarkers | 2-year
Quality of life | 2-year
  D15 questionnaire.
cognitive function | 2-year
  MMSE questionnaire
depressive symptoms | 2-year
  WHO-MINI questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Gabriel, MD, PhD, Principal Investigator — Evidem Consultores SL; Jaakko Tuomilehto, MD, PhD, Principal Investigator — Evidem Consultores SL
Locations (1):
- Centro de Salud Jose Marva, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Damanawi R, Stanley IK, Staatz C, Pascoe EM, Craig JC, Johnson DW, Mallett AJ, Hawley CM, Milanzi E, Hiemstra TF, Viecelli AK. Metformin for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2024 Jun 4;6(6):CD013414. doi: 10.1002/14651858.CD013414.pub2. PMID 38837240
- [Derived] Gabriel R, Boukichou Abdelkader N, Acosta T, Gilis-Januszewska A, Gomez-Huelgas R, Makrilakis K, Kamenov Z, Paulweber B, Satman I, Djordjevic P, Alkandari A, Mitrakou A, Lalic N, Colagiuri S, Lindstrom J, Egido J, Natali A, Pastor JC, Teuschl Y, Lind M, Silva L, Lopez-Ridaura R, Tuomilehto J; e-PREDICE Consortium. Early prevention of diabetes microvascular complications in people with hyperglycaemia in Europe. ePREDICE randomized trial. Study protocol, recruitment and selected baseline data. PLoS One. 2020 Apr 13;15(4):e0231196. doi: 10.1371/journal.pone.0231196. eCollection 2020. PMID 32282852
- See also: Webpage ePREDICE Project — http://www.epredice.eu
- Available data/document: Study Protocol — http://www.epredice.eu — Study Protocol Version 5.0